CLINICAL TRIAL: NCT02742571
Title: Validation of PINI Score in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0258
Record Dates: First submitted 2016-03-03; First posted 2016-04-19 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: ICU Patients
Keywords: Biological evaluation of denutrition; Denutrition; PINI score

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: non applicable

SUMMARY:
Prospective, observational clinical monocentric study in ICU; Relationship between Pronostic Inflammatory and Nutritional Index (PINI) (and biomarkers related to PINI) and mortality, morbidity and nutrition in ICU

DETAILED DESCRIPTION:
Main objective: to evaluate the relationship between PINI score and biomarker related to PINI, and 28 days mortality in ICU

Secondary objectives:

* to evaluate the relationship between PINI score (and biomarkers related to PINI) and morbidity in ICU : SOFA score, duration of ventilation, duration of antibiotherapy, duration of extra renal epuration, length of stay
* to evaluate the relationship between PINI score (and biomarkers related to PINI) and nutrition in ICU (type of nutrition, calorie content)

ELIGIBILITY:
Inclusion Criteria:

* Both patient in ICU

Exclusion Criteria:

* minor patient
* No possibility to calculate PINI score
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
PINI Score | at day 1
Biomarkers related to PINI | at day 1
Mortality at 28 days | after admission

SECONDARY OUTCOMES:
Length of stay | at day 1
Duration of ventilation | at day 1
Duration of antibiotherapy | at day 1
Duration of renal replacement therapy | at day 1
Type of nutrition (enteral/parenteral) | at day 1
Calorie content per day | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France